CLINICAL TRIAL: NCT03236090
Title: Study of the Effect of Vivomixx® on Neuroinflammation Ans Systemic Inflammatory Response in Patients With Cirrhosis
Brief Title: Effect of Vivomixx® on Neuroinflammation in Patients Withs Cirrhosis
Status: Withdrawn | Phase: Not Applicable | Type: Interventional
Why Stopped: Problems to recruit patients due to exclusion criteria
Sponsor: Fundació Institut de Recerca de l'Hospital de la Santa Creu i Sant Pau (Other)
Collaborators: Spanish Clinical Research Network - SCReN (Network)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: IIBSP-VIV-2016-109
Record Dates: First submitted 2017-06-29; First posted 2017-08-01 (Actual); Last update posted 2018-03-13 (Actual); Status verified 2018-03

CONDITIONS: Cirrhosis, Liver
Keywords: Cirrhosis; Probiotics; Systemic inflammation; neuroinflammation; Cognitive function; Bacterial translocation
MeSH Terms: conditions — Liver Cirrhosis; Fibrosis; Neuroinflammatory Diseases

STUDY DESIGN:
Intervention Model Description: Decompensated patients with cirrhosis:
  1. Outpatients with refractory ascites (substudy 1) (n=20)
  2. Patients hospitalized because bacterial infection (substudy 2) (n=30)
Who Masked: Participant
Masking Description: Placebo (we evaluate the probiotic Vivomixx® vs placebo as adjunctive in addition to the standard of care)
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Outpatients with refractory ascites (Active Comparator): 20 consecutive outpatients with cirrhosis and refractory ascites Vivomixx®sachets containing 450 x 109 bacteria, 2 every 12 hours (n=25), or placebo (n=25)
  Interventions: Dietary Supplement: Vivomixx
- Patients hospitalized because bacterial infection (Active Comparator): 30 consecutive patients with cirrhosis and bacterial infections. All patients will receive endovenous antibiotics and, only in the case of patients with SBP, also intravenous albumin Vivomixx®sachets containing 450 x 109 bacteria, 2 every 12 hours (n=25), or placebo (n=25)
  Interventions: Dietary Supplement: Vivomixx

INTERVENTIONS:
Dietary Supplement: Vivomixx — Vivomixx®sachets containing 450 x 109 bacteria, 2 every 12 hours (n=25), or placebo (n=25)

SUMMARY:
Study Design:

Double-blind randomized placebo-controlled clinical trial

Study Duration:

2 years

Study Center:

Single center Hospital de la Santa Creu i Sant Pau, Barcelona

Objectives:

To assess the effect of Vivomixx® on neuroinflammation and systemic inflammatory response in patients with cirrhosis

DETAILED DESCRIPTION:
Study variables Main variables

* Neuroinflammation
* Systemic inflammatory response Secondary variables
* Cognitive function
* Bacterial translocation
* Intestinal barrier
* Systemic oxidative damage
* Time until SBP or other bacterial infection resolution in patients with infections
* Incidence of complications of cirrhosis and mortality during the study 40 patients, 20 and 30 in each of the two substudies, respectively Diagnosis and Main Inclusion Criteria
* Decompensated patients with cirrhosis:

  1. Outpatients with refractory ascites (substudy 1) (n=20)
  2. Patients hospitalized because bacterial infection (substudy 2) (n=30)

Study Product:

Vivomixx®sachets containing 450 x 109 bacteria, 2 every 12 hours (n=25), or placebo (n=25)

Duration of administration:

30 days Follow up The following patients' assessments will be performed: in substudy 1 at baseline and at the end of the treatment (30 days), and in substudy 2 at baseline, on day 1, day 2, day 3, day 7, at infection resolution, and at discharge or day 30.

Clinical and analytical assessments will be performed every three months after the end of the study Comparator Placebo (we evaluate the probiotic Vivomixx® vs placebo as adjunctive in addition to the standard of care) Statistical Methodology Fisher's exact test for categorical variables and Student's "t" test and Mann-Whitney and Wilcoxon tests for quantitative variables. Correlations will be assessed by Spearman test. A two-sided p value <0.05 will be considered statistically significant

ELIGIBILITY:
Inclusion Criteria:

* Outpatients with cirrhosis and refractory ascites according to current definition (29) (substudy 1), and hospitalized patients with cirrhosis and an episode of bacterial infection (substudy 2) at Hospital de la Santa Creu i Sant Pau.

Cirrhosis will be diagnosed by clinical, analytical and ultrasonographic findings or by liver biopsy. SBP will be diagnosed by an ascitic fluid neutrophil count > 250/mm3 with or without positive culture (28). Bacteremia, urinary infections, pneumonia, cellulitis, other bacterial infections and possible or suspected infections will be diagnosed according to current guidelines (13,14,28). All patients with SBP, bacteremia or pneumonia will be included. However patients with urinary infections, cellulitis or suspected infection these non-SBP infections will be required to fulfil the following requirements: at least two criteria of SIRS (systemic inflammatory response syndrome) (Annex I) (30) and CRP (C-reactive protein) >= 10 mg/dl (28).

Exclusion Criteria:

* Advanced hepatocellular carcinoma (beyond Milan's criteria) or any other malignancy determining a poor short-term prognosis.
* Advanced liver insufficiency [MELD (model for end-stage liver disease) >25].
* Marked symptomatic comorbidities (neurological, cardiac, pulmonary, renal, psychiatric, HIV infection).
* Septic shock, ileus, need for tracheal intubation or intensive care unit.
* Immunomodulatory drugs.
* In substudy 1, any infection at inclusion in the study.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 0 (Actual)
Dates: Start 2017-07-15 (Actual); Primary Completion 2018-03-09 (Actual); Study Completion 2018-03-09 (Actual)

PRIMARY OUTCOMES:
Change in neuroinflammation | Change from baseline at 30 days
  For substudy 1, neuroinflammation will be measured by MRI at baseline and 30 days
Change in neuroinflammation | Change from baseline at 3 days
  For substudy 2, neuroinflammation will be measured by MRI at baseline and 3 days

CONTACTS AND LOCATIONS:
Locations (1):
- Hospital de la Santa Creu i Sant Pau, Barcelona, Spain

IPD SHARING:
Plan to Share IPD: No